CLINICAL TRIAL: NCT07272811
Title: Neurocognitive Assessment Platform 4 Alzheimer
Acronym: NAP4A2020
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Prof. Massimo Filippi, Prof., IRCCS San Raffaele
Other Study IDs: NAP4A2020
Record Dates: First submitted 2025-11-26; First posted 2025-12-09 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: MCI; MCI Conversion to Dementia; AMCI - Amnestic Mild Cognitive Impairment; Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- aMCI patients: Individuals diagnosed with single- or multi-domain amnestic MCI (aMCI)
- Healthy Controls: Healthy individuals (with similar sex, age, and education level to the aMCI group)

SUMMARY:
The aging population in Europe is leading to an increase in neurodegenerative diseases, such as Alzheimer's disease (AD), which is expected to affect 152 million people worldwide by 2050. In Italy, there are approximately 1.2 million cases of dementia, with 600,000 attributed to AD. Given the limited effectiveness of current pharmacological treatments, there is a growing need for early, non-pharmacological interventions to slow disease progression and improve the quality of life for patients and caregivers.

The Neurocognitive Assessment Platform 4 Alzheimer (NAP4A) study aims to create a digital platform for the early detection of amnestic mild cognitive impairment (MCIa), considered an intermediate stage between normal aging and dementia. The platform uses non-invasive biometric tools, including EEG, blood flow sensors, and eye-tracking devices, to collect neurophysiological and behavioral data.

The study will involve 100 participants aged 55 to 80, divided into two groups: one with individuals diagnosed with MCIa and a control group of healthy participants. Over 12 months, regular assessments will be conducted to identify markers that predict the progression from MCIa to AD. The goal is to develop advanced diagnostic tools that support early and targeted interventions.

ELIGIBILITY:
Inclusion criteria common to both experimental groups:

* Signature of informed consent
* Age between 55 and 80 years
* Absence of functional impact on daily living activities or minimal impact on instrumental activities

Specfic inclusion criteria for Healthy Controls recruitment:

* Normal global cognitive efficiency (Mini Mental State Examination scores of 28 or higher)
* Absence of specific cognitive deficits (memory and other cognitive domains) that are abnormal for age, sex, and education level (1.5 standard deviations below the mean for age- and education-matched controls), as assessed by objective, standardized cognitive tests.

Specific inclusion criteria for aMCI recruitment:

* Cognitive difficulties reported by the individual, their family member, or their primary care physician
* Normal global cognitive efficiency (Mini Mental State Examination score within 0.5 standard deviations of the average for age- and education-matched control subjects).
* Specific cognitive deficits related to memory or multi-domain cognitive impairments (involving memory and other cognitive domains) that are atypical for the individual's age (1.5 standard deviations below the average for age- and education-matched controls), as determined by objective, standardized cognitive tests.

Exclusion Criteria:

* Rejection of informed consent
* Important sensory deficits (e.g., hearing loss or hypovisus)
* Current or previous history of psychiatric illness
* Current or previous degenerative pathology of the central nervous system (CNS)
* Presence of systemic diseases in anamnesis
* Presence of cerebrovascular events in anamnesis
* Use of alcohol or psychotropic substances in anamnesis

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will involve around 100 participants aged 55-80, including 50 with aMCI (single or multiple domain) and 50 healthy controls. Patients will be recruited from the Neurology Unit or dementia care clinics at IRCCS Ospedale San Raffaele. Healthy controls will be selected from the general population based on the study's inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-12-15 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Development of NAP4A Platform | 12 months
  To create a digital tool for fast and easy cognitive and behavioral assessment to examine the preclinical stage of Alzheimer's: Neurocognitive Assessment Platform 4 Alzheimer (NAP4A)

SECONDARY OUTCOMES:
Early diagnosis of aMCI at risk of conversion to AD | 12 months
  To identify aMCI individuals at an early stage who are at risk of progression to AD using the Neurocognitive Assessment Platform 4 Alzheimer (NAP4A)
Identify the main predictive markers | 12 months
  To develop probability markers that predict the likelihood of aMCI individuals converting to AD based on data from the Neurocognitve Assessment Platform 4 Alzheimer

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS San Raffele, Milan, Italy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zucchella C, Sinforiani E, Tamburin S, Federico A, Mantovani E, Bernini S, Casale R, Bartolo M. The Multidisciplinary Approach to Alzheimer's Disease and Dementia. A Narrative Review of Non-Pharmacological Treatment. Front Neurol. 2018 Dec 13;9:1058. doi: 10.3389/fneur.2018.01058. eCollection 2018. PMID 30619031
- [Background] Yankner BA, Lu T, Loerch P. The aging brain. Annu Rev Pathol. 2008;3:41-66. doi: 10.1146/annurev.pathmechdis.2.010506.092044. PMID 18039130
- [Background] Petersen RC, Morris JC. Mild cognitive impairment as a clinical entity and treatment target. Arch Neurol. 2005 Jul;62(7):1160-3; discussion 1167. doi: 10.1001/archneur.62.7.1160. No abstract available. PMID 16009779
- [Background] Bherer L. Cognitive plasticity in older adults: effects of cognitive training and physical exercise. Ann N Y Acad Sci. 2015 Mar;1337:1-6. doi: 10.1111/nyas.12682. PMID 25773610
- [Background] Albert MS, DeKosky ST, Dickson D, Dubois B, Feldman HH, Fox NC, Gamst A, Holtzman DM, Jagust WJ, Petersen RC, Snyder PJ, Carrillo MC, Thies B, Phelps CH. The diagnosis of mild cognitive impairment due to Alzheimer's disease: recommendations from the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease. Alzheimers Dement. 2011 May;7(3):270-9. doi: 10.1016/j.jalz.2011.03.008. Epub 2011 Apr 21. PMID 21514249
- [Background] Sun Z, van de Giessen M, Lelieveldt BP, Staring M. Detection of Conversion from Mild Cognitive Impairment to Alzheimer's Disease Using Longitudinal Brain MRI. Front Neuroinform. 2017 Feb 24;11:16. doi: 10.3389/fninf.2017.00016. eCollection 2017. PMID 28286479